CLINICAL TRIAL: NCT05204524
Title: A Phase II Study of Temozolomide for Injection Combined With Epirubicin in the First-line Treatment of Leiomyosarcoma
Brief Title: Temozolomide for Injection Combined With Epirubicin in First-line Treatment of Leiomyosarcoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, yihebali chi, Deputy chief physician of internal medicine, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21/313-2984
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma | interventions — Temozolomide; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjected arm (Experimental): temozolomide for injection (once a day, with a fixed dose of 200 mg (body surface area ≤1.7m2) or 300 mg (body surface area > 1.7 m2), for 5 days, with 21 days as a cycle) combined with epirubicin (60 mg/m2 21-day scheme).
  Temozolomide for injection, according to the requirements of GCP, the test drug should be sealed, kept away from light and kept at 2-8℃, with a valid period of 24 months.
  Interventions: Drug: Temozolomide for injection combined with epirubicin

INTERVENTIONS:
Drug: Temozolomide for injection combined with epirubicin — Temozolomide for injection, according to the requirements of GCP, the test drug should be sealed, kept away from light and kept at 2-8℃, with a valid period of 24 months.

SUMMARY:
This study is a single-center, prospective, one-arm clinical study, which is planned to be carried out in Cancer Hospital of Chinese Academy of Medical Sciences. The patients with locally advanced or metastatic leiomyosarcoma who are inoperable are enrolled, aiming at the effectiveness and safety of temozolomide for injection combined with epirubicin as the first-line treatment for advanced leiomyosarcoma.

DETAILED DESCRIPTION:
Sarcoma is a rare solid tumor, accounting for about the malignant tumors in adults. About 80% of sarcoma originated from soft tissue, and the remaining 20% originated from bone. In a word, soft tissue sarcoma consists of more than 50 different histological subtypes. Leiomyosarcoma is one of the most common soft tissue sarcomas, and its incidence is estimated to be between 10% and 20% in all newly diagnosed soft tissue sarcomas. Leiomyosarcoma accounts for a large proportion of soft tissue and abdominal-pelvic sarcoma, second only to liposarcoma, and is the main sarcoma caused by large vessels. In addition, uterine leiomyosarcoma mainly comes from smooth muscle cells in myometrium, which can exist alone or coexist with leiomyoma, and is the most common uterine sarcoma.

Local and distant metastasis can occur in leiomyosarcoma. Generally speaking, patients with leiomyosarcoma whose tumor diameter is less than 5cm have a better prognosis. More than 40% of dermal tumors are prone to recurrence, but rarely metastasize. On the contrary, 1/3 of subcutaneous tumors can metastasize, with poor prognosis, and often metastasize to liver and lung, which requires regular follow-up visits to hospitals. Leiomyosarcoma from skin has a good prognosis and can be cured. Leiomyosarcoma originating from soft tissues, bones and blood vessels of trunk has poor prognosis and generally cannot be completely cured.

Surgical resection is the main treatment for leiomyosarcoma, and the tumor tissue should be completely removed as far as possible. Those involved in lymph nodes which are within the scope of resection should be removed together, but lymph node dissection is not advocated. After operation, active chemotherapy and active prevention should be taken to prevent recurrence. The treatment period is 6 ~ 12 months. As an auxiliary treatment after surgery, radiotherapy is a non-invasive treatment. Preoperative radiotherapy can improve the resection rate and organ preservation rate, while postoperative radiotherapy can reduce the local recurrence rate and improve the survival rate.

The most life-threatening aspect of leiomyosarcoma is its tendency to blood-borne transmission, so it needs systemic control. For patients who cannot be completely removed after surgical resection or who will cause severe physical disability or even life-threatening. However, the treatment of resectable and metastatic diseases is still unsatisfactory because leiomyosarcoma is moderately sensitive to chemotherapy. Only three drugs-epirubicin, ifosfamide and dacarbazine (DTIC) have effective activity in patients with soft tissue sarcoma, and the response rate is about 20%3-4 in the second phase study. Compared with single drug, combined chemotherapy did not improve the overall survival rate by 4-6. The median survival rate was still about 12 months. Obviously, it is necessary to find new drugs with soft tissue sarcoma activity to improve the treatment of these tumor patients.

Temozolomide is an alkylating agent and an antitumor drug, which can pass through the blood-cerebrospinal fluid barrier and is clinically used for the first-line treatment of brain tumors. Cytotoxicity caused by DNA methylation and mismatch repair 6-7. A Phase II clinical study on the efficacy and toxicity of temozolomide in patients with unresectable or metastatic soft tissue sarcoma. Results The dosage regimen of temozolomide used in the study was well tolerated and had moderate activity against unresectable or metastatic leiomyosarcoma of uterus and non-uterus. In 25 patients, the overall objective remission rate was 8%. At the median follow-up of 13.2 months, the median progression-free survival time and median overall survival time were 2.0 months (95% confidence interval [95% CI], 1.7-2.3) and 13.2 months (95% CI, 4.7-31.1), respectively. All patients suffered from uterine leiomyosarcoma or non-uterine leiomyosarcoma. In the subset analysis of these patients, the objective remission rate was 18% (2 out of 11 patients), while the disease stabilized in 3 out of 11 patients (27%). For this subgroup, the median follow-up time was 24.4 months, the median progression-free survival time and median overall survival time were 3.9 months (95% CI, 1.9-21.9) and 30.8 months (lower limit 95% CI, 7.8), respectively.

A single dose of epirubicin is the standard systemic treatment for soft tissue sarcoma, followed by leiomyosarcoma. Epirubicin, as a single drug, has a reported response rate of 10% to 25% (Krikelis and Judson analyzed retrospectively in 2010), although leiomyosarcoma seems to be inferior to other sarcoma subtypes, such as synovial sarcoma and liposarcoma. Retrospective clinical data of 2185 patients with sarcoma treated with epirubicin showed that the response rate of leiomyosarcoma was low (11%).

Therefore, this study designed to evaluate the efficacy and safety of temozolomide for injection combined with epirubicin in the first-line treatment of advanced leiomyosarcoma, and to observe and evaluate the efficacy and safety of temozolomide for injection combined with epirubicin in the first-line treatment of advanced leiomyosarcoma.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients voluntarily participated in this study and signed informed consent; 2. Unresectable, locally advanced or metastatic leiomyosarcoma, and never received systemic treatment, including chemotherapy, targeted therapy and immunotherapy; 3.18~70 years old (including 18 and 70 years old), male or female. 4.ECOG PS score: 0~2 points; 5. The estimated survival time is more than 3 months; 6. The main organ function meets the following criteria within 7 days before treatment:

A. blood routine examination standard (without blood transfusion within 14 days):

* hemoglobin (HB) ≥ 90g/l; ② absolute neutrophil count (ANC) ≥ 1.5× 109/l; ③ platelet (PLT)≥80×109/L ..

B. biochemical examination shall meet the following standards:

* total bilirubin (TBIL)≤1.5 times the upper limit of normal value (uln);

  * Alanine aminotransferase (ALT) and aspartate aminotransferase AST≤2.5ULN, and ALT and AST ≤ 5 ULN with liver metastasis;

    * serum creatinine (Cr)≤1.5ULN or creatinine clearance rate (CCR) ≥ 55ml/min; C. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF)≥ the lower limit of normal value (50%).

      7. Women of childbearing age should agree that contraceptive measures (such as intrauterine device, contraceptive pill or condom) must be used during the study and within 6 months after the end of the study; Serum or urine pregnancy test was negative within 7 days before the study entered the group, and it must be a non-nursing patient. Men should agree to patients who must use contraception during the study period and within 6 months after the end of the study period.

      8. There must be at least one measurable lesion meeting the RECIST 1.1 standard (the measured diameter line shall be based on the longest diameter of the lesion ≥10mm, and the shortest diameter of lymph nodes ≥15mm).

Exclusion Criteria:

* 1.Or accompanied by other malignant tumors in the past, except the cured basal cell carcinoma of skin and carcinoma in situ of cervix; 2. Those who have been proved to be allergic to temozolomide, dacarbazine or DTIC, epirubicin and/or their auxiliary materials; 3. Special attention: Patients with gastrointestinal bleeding risk should not be included in the group, including the following situations: (1) Active peptic ulcer lesions with occult blood in stool (++); (2) Those who have a history of black stool and hematemesis within 3 months; (3) Gastroscopy must be performed for fecal occult blood (+) to determine whether organic diseases of gastrointestinal tract exist; 4. There were active heart diseases, including myocardial infarction, severe/unstable angina pectoris, etc. Echocardiographic left ventricular ejection fraction < 50% and poorly controlled arrhythmia (including QTcF interval > 450 ms for men and > 470ms)； for women); 5. Severe infection (such as intravenous drip of antibiotics, antifungal or antiviral drugs) occurred within 6 months before enrollment, or fever of unknown cause occurred during screening/before first administration > 38.5°C；; 6. Those with abnormal coagulation function (INR>1.5×ULN, APTT>1.5×ULN) and bleeding tendency; 7. Pregnant or lactating women; Prohibited in patients with severe myelosuppression; 8. The researcher believes that there are any conditions that may harm the subject or cause the subject to fail to meet or implement the research requirements; 10. Those who have a history of psychotropic drug abuse and cannot quit or have mental disorders; 11. According to the judgment of the researcher, there are accompanying diseases that seriously endanger the patient's safety or affect the patient's completion of the study;

Rejection study:

1. Failure to use drugs according to the provisions of this plan leads to failure to evaluate the effectiveness and/or safety;
2. In the course of research and treatment, researchers are allowed to give corresponding supportive treatment according to the clinical needs of subjects, and anti-tumor treatment not specified in the research scheme is prohibited in the course of treatment, but medical measures taken for tumor emergencies that endanger patients' lives are not included.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-08-27 (Estimated); Study Completion 2023-08-27 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 42 days
  The objective curative effect of tumor was evaluated by recist version 1.1 standard, including the percentage of patients with complete remission and partial remission maintained for more than 4 weeks.

SECONDARY OUTCOMES:
Disease control rate | 42 days
  Including complete remission, partial remission and stable disease, and the number of cases maintained for more than 4 weeks.
progression-free survival | 42 days
  The time from the first administration to the objective progression or death of tumor.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China